CLINICAL TRIAL: NCT03981289
Title: GRASP-LGMD: Defining Clinical Endpoints in LGMD
Brief Title: Defining Clinical Endpoints in Limb Girdle Muscular Dystrophy (LGMD)
Acronym: GRASP-01-001
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Newcastle University (Other); Nationwide Children's Hospital (Other); Washington University School of Medicine (Other); University of Iowa (Other); University of Minnesota (Other); University of California, Irvine (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); University of Colorado, Denver (Other); University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HM20018721; GRASP-LGMD (Other: Virginia Commonwealth University)
Record Dates: First submitted 2019-06-03; First posted 2019-06-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Limb Girdle Muscular Dystrophy; Muscular Dystrophies
Keywords: LGMD; Limb Girdle Muscular Dystrophy; CAPN3; ANO5; DYSF; DNAJB6; Sarcoglycan; SGCA; SGCB; SGCD; SGCG
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Muscular Dystrophies; Muscular Dystrophy, Limb-Girdle, Type 1D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- CAPN3 (LGMD2A): Clinical Assessments, Biomarkers
- DYSF (LGMD2B): Clinical Assessments, Biomarkers
- ANO5 (LGMD2L): Clinical Assessments, Biomarkers
- DNAJB6 (LGMD1D): Clinical Assessments, Biomarkers
- Sarcoglycan (LGMD2D) (LGMD2E) (LGMD2C) (LGMD2F): Clinical assessments

SUMMARY:
Limb Girdle Muscular Dystrophy comprise a group of disorders made up of over 30 mutations which share a common phenotype of progressive weakness of the shoulder and hip girdle muscles. While the individual genetic mutations are rare, as a cohort, LGMDs are one of the four most common muscular dystrophies. The overall goal of project 1 is to define the key phenotypes as measured by standard clinical outcome assessments (COAs) for limb girdle muscular dystrophies (LGMD) to hasten therapeutic development.

DETAILED DESCRIPTION:
The genetic heterogeneity has been a barrier to broad natural history efforts, with prior investigations often limited to single gene mutations. Much attention is paid to the variability within individual mutations (e.g. distal presentations), as opposed to defining the best strategy for measuring change in overall LGMD disease burden. This presents a major dilemma for LGMD rare disease research: how to balance diverse genes leading to overlapping phenotypes, versus variants in the same gene leading to divergent phenotypes. What is clear, is as a group, LGMDs are chronic and progressive leading to significant lifetime morbidity and represent a large unmet clinical need.

Recent developments in the investigator's genetic understanding of LGMD and molecular approaches to therapy have led to proposed gene replacement therapies for at least three of the LGMD mutations. Several of these gene replacement therapies are currently in pre-clinical/phase 1 testing, leading to an urgent need for natural history data. In addition, non-specific therapies which target muscle mass or function are being tested in other muscular dystrophies and may prove beneficial for LGMD.

ELIGIBILITY:
Inclusion Criteria - Arm 1:

* Age between 4-65 at enrollment
* Clinically affected (defined as weakness on bedside evaluation in either a limb-girdle pattern, or in a distal extremity)
* A genetically or functionally confirmed mutation in ANO5, CAPN3, DYSF, DNAJB6 or SGCA-G.
* Willing and able to give informed consent and follow all study procedures and requirements

Inclusion Criteria - Arm 2:

* Age between 4-65 at enrollment
* Clinically affected (defined as weakness on bedside evaluation in either a limb-girdle pattern, or in a distal extremity)
* a genetically confirmed mutation in SGCA-G
* Willing and able to give informed consent and follow all study procedures and requirements

Exclusion Criteria - Arm 1:

* Any other illness that would interfere with the ability to undergo safe testing or would interfere with interpretation of the results in the opinion of the site investigator.
* History of a bleeding disorder, platelet count <50,000, current use of an anticoagulant.
* Positive pregnancy test at time any timepoint during the trial.

Exclusion Criteria - Arm 2:

* Any other illness that would interfere with the ability to undergo safe testing or would interfere with interpretation of the results in the opinion of the site investigator.
* History of a bleeding disorder, platelet count <50,000, current use of an anticoagulant
* Positive pregnancy test at time any timepoint during the trial.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GRASP-LGMD covers a broad geographical distribution and we expect the race and ethnicity to match that of the United States. However, past experience in both the clinical and research LGMD populations shows that some minority subgroups are under-represented in research studies. To assist with recruitment of persons from diverse backgrounds we will utilize the Community and Special Populations Engagement Personnel supported through the CTSA networks to reach out to under-represented communities through a variety of local techniques which could include direct outreach, advertising with local advocacy groups, organizations, or newsletters, and local advertising using a variety of media which could include Social Media (e.g. Facebook, Twitter), radio, and newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mobility | Baseline to 12 months
  Mobility will be measured using the 100 Meter Timed Test (100m) in which the participant is asked to complete 2 laps around 2 cones set 25 meters apart as quickly as safely possible, running if able, and the time in seconds is recorded.
Change in motor performance | Baseline to 12 months
  The North Star Assessment for Dysferlinopathy (NSAD) is a functional scale specifically designed to measure motor performance in individuals with LGMD. It consists of 29 items that are considered clinically relevant items from the North Star Ambulatory Assessment and the Motor Function Measure 20 with a maximum score of 54 and higher scores indicate higher functional abilities.
Change in upper limb function characteristics | Baseline to 12 months
  The Performance of Upper Limb 2.0 (PUL) scale measures the progression of weakness and natural history of functional decline in Duchenne muscular dystrophy. There are 22 scored items; a score of 42 indicates the highest level of independent function and 0 the lowest.
Change in Forced vital capacity (FVC) | Baseline to 12 months
  Volume of air forcefully exhaled will be measured using Spirometry performed in a sitting position using standardized equipment
Changes in Forced expiratory volume (FEV1) | Baseline to 12 months
  Volume of air forcefully exhaled in one second will be measured using Spirometry performed in a sitting position using standardized equipment
Change in activity limitations | Baseline to 12 months
  ACTIVLIM is a patient-reported measure of activity limitations for individuals with upper and/or lower limb impairments, which measures the ability to perform daily activities.
Change in self-reported physical health | Baseline to 12 months
  PROMIS Physical Health is part of a set of patient-reported measures developed by a National Institute of Health that evaluates general physical health by assessing fatigue, pain intensity, pain interference, physical function, sleep disturbance, dyspnea, gastrointestinal symptoms, itch, pain behavior, pain quality, sexual function, and sleep related impairment.
Change in overall health | Baseline to 12 months
  Domain Delta Questionnaire is a patient reported measure that assesses overall health over the previous 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (10):
- United States (9):
  - University of California Irvine, Irvine, California
  - The University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
- John Walton Muscular Dystrophy Research Centre (Newcastle Upon Tyne), Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated and deidentified data will be shared with qualified investigators upon majority approval of the LGMD investigators

REFERENCES:
- [Derived] Doody A, Alfano L, Diaz-Manera J, Lowes L, Mozaffar T, Mathews KD, Weihl CC, Wicklund M, Hung M, Statland J, Johnson NE; GRASP-LGMD Consortium. Defining clinical endpoints in limb girdle muscular dystrophy: a GRASP-LGMD study. BMC Neurol. 2024 Mar 15;24(1):96. doi: 10.1186/s12883-024-03588-1. PMID 38491364
- [Derived] Doody A, Alfano L, Diaz-Manera J, Lowes L, Mozaffar T, Mathews K, Weihl CC, Wicklund M, Statland J, Johnson NE; GRASP-LGMD Consortium. Defining Clinical Endpoints in Limb Girdle Muscular Dystrophy: A GRASP-LGMD study. Res Sq [Preprint]. 2023 Oct 6:rs.3.rs-3370395. doi: 10.21203/rs.3.rs-3370395/v1. PMID 37886601